CLINICAL TRIAL: NCT03166579
Title: Evaluating the Effectiveness of 'The Endeavour Programme': DBT for Irish Adults With Borderline Personality Disorder
Brief Title: Effectiveness Evaluation of 'The Endeavour Programme'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Mary Joyce, Project Co-ordinator, Health Service Executive, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOSP
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Personality Disorder, Borderline
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dialectical Behaviour Therapy (Experimental): Participants receive the "standard" 12 month DBT programme where all four modes of treatment are delivered including: individual therapy, group skills training, telephone coaching and DBT team consultation.
  Interventions: Behavioral: Dialectical Behaviour Therapy

INTERVENTIONS:
Behavioral: Dialectical Behaviour Therapy — Dialectical Behaviour Therapy (DBT) is a psychological intervention which was originally developed for women with Borderline Personality Disorder. DBT is delivered by a team of multidisciplinary mental health professionals, and comprises of individual therapy sessions for each patient, group skills training sessions, phone coaching and consultation meetings for the clinicians on the DBT team. Group skills are delivered in blocks of three modules which teach mindfulness, distress tolerance, emotion regulation and interpersonal effectiveness. The three modules are delivered over a 24-week period and are then repeated.

SUMMARY:
This study aims to evaluate the effectiveness of Dialectical Behaviour Therapy for adults with Borderline Personality Disorder attending Community Mental Health Services in Cork, Ireland.

The main objective of the current study is to determine if completion of a 12 month DBT programme is associated with improved outcomes in terms of borderline symptoms, anxiety, hopelessness, suicidal behaviour, depression and quality of life.

A secondary objective includes assessing client progress across multiple time-points throughout the treatment.

DETAILED DESCRIPTION:
Dialectical Behaviour Therapy (DBT) is noted to be an intervention with a growing evidence base which demonstrates its effectiveness in treating individuals with Borderline Personality Disorder (BPD). Nine randomised controlled trials have been completed at six independent sites. These trials have found a reduction in suicidal behaviours, intentional self-injury, depression, hopelessness and other difficulties associated with this mental health diagnosis.

While the efficacy of DBT has been demonstrated through multiple RCTs, few studies have examined the effectiveness of DBT in community mental health settings. In particular, no study to our knowledge has evaluated the standard 12-month DBT programme for adults with BPD in an Irish community setting. "Standard" DBT is delivered by a team of multidisciplinary mental health professionals, and comprises of individual therapy sessions for each patient, group skills training sessions, phone coaching and consultation meetings for the clinicians on the DBT team.

The current study thus aims to evaluate the effectiveness of the standard 12-month DBT programme (The Endeavour Programme) in an Irish community setting.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for diagnosis of either Borderline Personality Disorder (DSM IV/V) or Emotionally Unstable Personality Disorder (ICD-10)
* Current emotion and behavioural dysregulation
* A history of self-harm behaviour
* The client will have discussed the diagnosis with a member of the DBT team and will have expressed an interest in, and commitment to the 12 month programme.

Exclusion Criteria:

* An active psychosis
* If the client has severe developmental delays, cognitive impairment or learning disabilities (exceeding mild range)
* If a clients' substance/drug dependence, eating disorder or any other mental health issue/behaviour is at such a level that it would impede their engaging with any of the modalities of DBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Borderline Symptoms | 12 months from pre-intervention to post-intervention
  Borderline Symptom List (BSL-23). The BSL-23 is a self-report questionnaire which comprises 23 items measuring borderline-typical symptomatology.
Suicidal ideation | 12 months from pre-intervention to post-intervention
  Beck Scale for Suicide Ideation (BSS). The BSS is a 21-item self-report assessment developed to identify individuals at risk of suicide.
Hopelessness | 12 months from pre-intervention to post-intervention
  Beck Hopelessness Scale (BHS). The BHS is a 20 item self-report measure which assesses key aspects of hopelessness.
Depression | 12 months from pre-intervention to post-intervention
  Beck Depression Inventory - Second Edition (BDI-II). The BDI-II is a 21 item self-report measure of symptoms and attitudes related to depression.
Anxiety | 12 months from pre-intervention to post-intervention
  Beck Anxiety Inventory (BAI). The BAI is a 21 is self-report multiple choice survey which evaluates both physiological and cognitive symptoms of anxiety
Quality of Life | 12 months from pre-intervention to post-intervention
  World Health Organisation Quality of Life Questionnaire (WHOQOL-BREF). The WHOQOL-BREF was developed collaboratively in a number of centres to act as an international cross-culturally comparable quality of life assessment. It comprises 26 items across four domains: physical health (domain 1), psychological health (domain 2), social relationships (domain 3), and environment (domain 4).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Flynn, PGDip, Principal Investigator — Psychology Manager

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flynn D, Kells M, Joyce M, Corcoran P, Gillespie C, Suarez C, Weihrauch M, Cotter P. Standard 12 month dialectical behaviour therapy for adults with borderline personality disorder in a public community mental health setting. Borderline Personal Disord Emot Dysregul. 2017 Sep 23;4:19. doi: 10.1186/s40479-017-0070-8. eCollection 2017. PMID 28989706